CLINICAL TRIAL: NCT00752544
Title: Phase I, Double-blind, Randomized, Placebo-controlled Trial to Examine the Safety, Tolerability and Plasma Pharmacokinetics of Ascending Oral Doses of TMC435350 After Single and Repeated Dosing in Healthy Japanese Male Subjects
Brief Title: TMC435350-TiDP16-C109: A Safety Study for TMC435350 in an Oral Solution Containing Either 100, 200 or 400 mg Equivalent of TMC435350 or Placebo in Healthy Japanese Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CR015418
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: HCV
Keywords: TMC435350; HCV; Hepatitis C; TMC435350-TiDP16-C109; TMC435350-C109
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir

INTERVENTIONS:
Drug: TMC435350

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of three different doses of TMC435350 compared to placebo in healthy Japanese males.

DETAILED DESCRIPTION:
This is a Phase I, double-blind (neither the physician or the volunteer knows the dose of the study medication), randomized (study medication assigned by chance), placebo-controlled (dose without the study medication present) trial to determine the safety, tolerability and plasma pharmacokinetics (amount of medication in the blood) of TMC435350 after single and multiple oral doses in healthy male Japanese volunteers. 100 mg, 200 mg and 400 mg doses will be given as an oral solution. Six (6) doses will be given with a 3 day follow-up between the first and second dose. Additional follow-up will be done for 3 days after the last dose and at approximately 2 and 4 weeks after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male volunteers between the ages of 20 and 55 years
* Japanese healthy volunteers who have resided outside of Japan for no more than five years and whose parents and maternal and paternal grandparents are Japanese
* Non-smoking or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months prior to selection
* Normal weight as defined by a Body Mass Index (BMI: weight in kg divided by square of height in meters) of 18.0 to 30.0 kg/m2
* Body weight above 50 kg at screening
* Informed Consent Form (ICF) signed voluntarily before any trial-related activity
* Normal 12-lead electrocardiogram (ECG) at screening
* Healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality.

Exclusion Criteria:

* Healthy volunteers must not have any of the following characteristics: Past history of heart arrhythmias (extrasystoli, tachycardia at rest) or having baseline prolongation of QTc interval > 450 ms, history of risk factors for Torsade de Pointes syndrome (hypokalemia, hypomagnesemia, family history of long QT Syndrome) or echographically suspected cardiomyopathy
* History or evidence of current use of alcohol, barbiturate, amphetamine, recreational or narcotic drug use which in the investigator's opinion would compromise healthy volunteer's safety and/or compliance with the trial procedures
* Hepatitis A, B, or C infection (confirmed by hepatitis A antibody, hepatitis B surface antigen, or hepatitis C virus antibody, respectively) or human immunodeficiency virus - type 1 (HIV-1) or HIV-2 infection at screening
* A positive urine drug test at screening. Urine will be tested for the presence of amphetamines, benzodiazepines, cocaine, cannabinoids, and opioids
* Currently active or underlying gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory, or infectious disease
* Any history of clinically relevant skin disease such as, but not limited to, dermatitis, eczema, drug rash, drug allergy, psoriasis, food allergy, urticaria
* History of drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy
* Use of concomitant medication, including herbal medications and dietary supplements and products containing Hypericum perforatum (e.g. St. John's wort), except for paracetamol (acetaminophen) or ibuprofen in a period of 14 days before the first trial medication intake
* Participation in another investigational drug trial within 30 days prior to the first intake of trial medication
* Donation of blood or plasma within 60 days preceding the first intake of trial medication

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Determine the short-term safety and tolerability of TMC435350 in healthy Japanese male volunteers after single and multiple doses and determine the plasma pharmacokinetics of TMC435350 after single and multiple doses.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Limited Clinical Trial, Study Director — Tibotec Pharmaceutical Limited